CLINICAL TRIAL: NCT06213220
Title: A Diagnostic Test of Mood Disorder Recognition in Children and Adolescents Based on Wearable Devices
Brief Title: Wearable Devices System Diagnoses Mood Disorder in Children and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Psychology, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: E2KM011639-MDCA
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-11

CONDITIONS: Mood Disorders; Diagnosis, Psychiatric
MeSH Terms: conditions — Mood Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mood disorders group: Participants are requested to wear the wristbands throughout the experiment, and upload their data every three days. Additionally, the Hamilton Depression Rating Scale (HAMD) and the Young Mania Rating Scale (YMRS) are administered once a week for measurement.
- healthy control group: Participants are requested to wear the wristbands throughout the experiment, and upload their data every three days. Additionally, the Hamilton Depression Rating Scale (HAMD) and the Young Mania Rating Scale (YMRS) are administered once a week for measurement.

SUMMARY:
As a diagnostic test, this study aims to explore the effectiveness of systems based on wearable devices in identifying mood disorders in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the MDD group met the DSM-5 diagnostic criteria for MDD and those in the BD group met the DSM-5 criteria for BD
* able to cooperate to complete the study
* had signed the informed consent prior to the study

Exclusion Criteria:

* with severe physical illness
* demonstrated symptoms comorbid with other psychiatric disorders (e.g., schizophrenia, conduct disorder, personality disorder) and developmental disorders (e.g., autism spectrum disorder, intellectual impairment)
* other conditions deemed inappropriate for inclusion in the group

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children and adolescents mood disorders patients and healthy controls age between 6 - 16 boys and girls
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
R-R interval | In the experiment conducted over a period of four weeks, the sampling frequency was 25Hz (based on seconds).The report will be available approximately one year after the end of the experiment.
  the interval between heart beats derived from Photoplethysmography (PPG)
Hamilton Depression Rating Scale (HAM-D) | In the experiment conducted over a period of four weeks, data collection was performed once per week. The report will be available approximately one year after the end of the experiment.
  Hamilton Depression Rating Scale (HAM-D) is the most widely used clinician-administered depression assessment scale. The original HAM-D has 21 items, but scoring is based only on the first 17. The patient is rated by a clinician on 17 items scored on a 5-point Likert-type scale. The total score ranges from 0 to 68. A score of 0-7 is considered to be normal while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.
Young Mania Rating Scale (YMRS) | In the experiment conducted over a period of four weeks, data collection was performed once per week. The report will be available approximately one year after the end of the experiment.
  The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. Additional information is based upon clinical observations made during the course of the clinical interview. The items are selected based upon published descriptions of the core symptoms of mania. The YMRS follows the style of the Hamilton Rating Scale for Depression (HAM-D) with each item given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Here's a quick list of what each score range may indicate in a patient: Less than or equal to 12 = remission; 13 -19 = minimal symptoms; 20 - 25 = mild mania; 26 - 37 = moderate mania; 38 - 60 = severe mania

OTHER OUTCOMES:
sensitivity | The model fitting will be completed approximately 6 months after the end of the experiment. The report will be available approximately one year after the end of the experiment.
  TP/(TP + FN) = (Number of true positive assessment)/(Number of all positive assessment) It measures the performance of the predictive model based on the primary outcome.
specificity | The model fitting will be completed approximately 6 months after the end of the experiment. The report will be available approximately one year after the end of the experiment.
  TN/(TN + FP) = (Number of true negative assessment)/(Number of all negative assessment) It measures the performance of the predictive model based on the primary outcome.
accuracy | The model fitting will be completed approximately 6 months after the end of the experiment. The report will be available approximately one year after the end of the experiment.
  (TN + TP)/(TN+TP+FN+FP) = (Number of correct assessments)/Number of all assessments) It measures the performance of the predictive model based on the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychology, Chinese Academy of Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No